CLINICAL TRIAL: NCT04247854
Title: Probiotic Bacillus for Decolonization of Methicillin-resistant Staphylococcus Aureus (MRSA) in Patients Undergoing Total Joint Arthroplasty: A Randomized, Prospective, Placebo-Controlled Pilot Study
Brief Title: Probiotics Pilot Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-01 JP
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Staphylococcus Aureus
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Bacillus subtilis probiotic
- No intervention (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis probiotic — Bacillus probiotic which contains one confidential ingredient of Bacillus subtilis spores (2 x 1010 CFU/g). Over 5 days of interventional period, the patient receives one tablet (250 mg; 5 x 109 CFU) of probiotic per day.
  Arms: Probiotic
Other: Placebo — Over 5 days of interventional period, the patient receives 1 placebo tablet per day
  Arms: No intervention

SUMMARY:
This pilot study is designed to determine if ingestion of Bacillus probiotics can cause alteration in levels of S. aureus colonization in the nose and intestine in preoperative orthopedic patients undergoing elective primary TJA.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age >18 years)
2. Undergoing elective primary knee or hip arthroplasty
3. Confirmed colonization of nares and/or rectum with S. aureus or MRSA on routine standard-of-care preadmission testing
4. Written informed consent

Exclusion Criteria:

1. Regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment
2. Antibiotic use within 3 months prior to enrollment
3. Active clinical infection
4. Participation in other clinical trials
5. Presence of pregnancy or lactation

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-01-22 (Estimated); Study Completion 2021-01-22 (Estimated)

PRIMARY OUTCOMES:
Persistent Staphylococcus aureus colonization | post-intervention: following 5 days of dietary supplementation

SECONDARY OUTCOMES:
Changes in microbiome composition | post-intervention: following 5 days of dietary supplementation
  as determine through next generation sequencing of samples collect from the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States